CLINICAL TRIAL: NCT05040373
Title: Patisiran-LNP Pregnancy Surveillance Program
Brief Title: Patisiran-Lipid Nanoparticle (LNP) Pregnancy Surveillance Program
Status: Recruiting | Type: Observational
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-TTR02-010
Record Dates: First submitted 2021-07-14; First posted 2021-09-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Transthyretin-mediated (hATTR) Amyloidosis; Polyneuropathy
Keywords: Hereditary neuropathic amyloidosis; Familial amyloidosis; Amyloidosis; Amyloidosis senile; Cardiac amyloidosis
MeSH Terms: conditions — Amyloidosis; Polyneuropathies; Amyloid Neuropathies, Familial; Amyloidosis, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patisiran: Pregnant women exposed to commercial patisiran-LNP (ONPATTRO) during the 12 weeks prior to their last menstrual period (LMP) or at any time during pregnancy.

SUMMARY:
The purpose of this study is to collect and evaluate pregnancy outcomes, pregnancy complications, and fetal/neonatal/infant outcomes in women exposed to patisiran-LNP.

ELIGIBILITY:
Inclusion Criteria:

* Documentation that the patient was exposed to patisiran-LNP at any point starting from 12 weeks before LMP or at any point during pregnancy

Exclusion Criteria:

* There are no exclusion criteria for participation in this program.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any woman exposed to patisiran-LNP 12 weeks prior to their last menstrual period (LMP) or at any time during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2030-10-12 (Estimated); Study Completion 2030-10-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Major Congenital Malformations | From 12 weeks prior to last dose of patisiran through one year after birth (Up to 21 months)
  Major congenital malformations will be classified according to the European Concerted Action on Congenital Anomalies and Twins (EUROCAT) and Metropolitan Atlanta Congenital Defects Program (MACDP) classification systems.

SECONDARY OUTCOMES:
Prevalence of Minor Congenital Malformations | From 12 weeks prior to last dose of patisiran through one year after birth (Up to 21 months)
  Minor congenital malformations will be classified classified according to the EUROCAT and MACDP classification systems.
Prevalence of Pregnancy Outcomes | From 12 weeks prior to last dose of patisiran through one year after birth (Up to 21 months)
  Pregnancy outcomes are defined as live birth, spontaneous abortions, stillbirths, elective abortions, molar or pregnancy, ectopic pregnancy, preterm births, and maternal death.
Prevalence of Other Adverse Fetal/Neonatal/Infant Outcomes | From 12 weeks prior to last dose of patisiran through one year after birth (Up to 21 months)
  Other adverse fetal/neonatal/infant outcomes are defined as low birth weight, failure to thrive, small for gestational age, postnatal growth and development, neonatal, and perinatal, or infant death.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (7):
- Clinical Trial Site, Iowa City, Iowa, United States
- Clinical Trial Site, Nantes, France
- Clinical Trial Site, Münster, Germany
- Clinical Trial Site, Pavia, Italy
- Clinical Trial Site, Groningen, Netherlands
- Clinical Trial Site, Lisbon, Portugal
- Clinical Trial Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No